CLINICAL TRIAL: NCT01318109
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of SYR-322 When Used in Combination With Metformin in Subjects With Type 2 Diabetes in Japan
Brief Title: Efficacy and Safety of Alogliptin Used Combination With Metformin in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322/CCT-006; JapicCTI-080629 (Registry Identifier: JapicCTI); UMIN000001394 (Registry Identifier: UMIN-CTR); U1111-1119-6303 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alogliptin 12.5 mg QD and metformin 500mg BID or 750mg TID (Active Comparator)
  Interventions: Drug: Alogliptin and metformin
- Alogliptin 25mg QD and metformin 500mg BID or 750mg TID (Active Comparator)
  Interventions: Drug: Alogliptin and metformin
- Metformin 500mg BID or 750mg TID (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Alogliptin and metformin — Alogliptin 12.5 mg, tablets, orally, once daily and metformin 250 mg, tablets, orally, twice or three times daily for up 12 weeks.
  Other Names: SYR-32; Glycoran
  Arms: Alogliptin 12.5 mg QD and metformin 500mg BID or 750mg TID
Drug: Alogliptin and metformin — Alogliptin 25 mg, tablets, orally, once daily and metformin 250 mg, tablets, orally, twice or three times daily for up 12 weeks.
  Other Names: SYR-322; Glycoran
  Arms: Alogliptin 25mg QD and metformin 500mg BID or 750mg TID
Drug: Metformin — Metformin 250 mg, tablets, orally, twice or three times daily and alogliptin placebo-matching tablets, orally, once daily for up 12 weeks.
  Other Names: Glycoran
  Arms: Metformin 500mg BID or 750mg TID

SUMMARY:
The purpose of this study was evaluate the efficacy and safety of alogliptin, once dairy (QD) combined with metformin taken twice daily (BID) or three times daily (TID) in type 2 diabetic patients with uncontrolled blood glucose.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

The present study was planned to evaluate the efficacy and safety of alogliptin as an add-on to metformin in type 2 diabetic patients who have uncontrolled blood glucose despite treatment with metformin as well as diet and exercise therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Had been taking metformin at a stable dose regimen (500 mg/day twice daily after meal or 750 mg/day three times daily after meal) for at least 12 weeks prior to the initiation of the treatment period (Week 0).
2. Had an glycosylated hemoglobin (HbA1c) of 6.5% or more and below 10.0% at 8 weeks after the initiation of the observation period (Week -4).
3. Had an HbA1c difference between 4 weeks after the initiation of the observation period (Week -8) and 8 weeks after the initiation of the observation period (Week -4) being within 10.0%* of the value at 4 weeks after the initiation of the observation period (Week -8) (*rounded off to the first decimal place).
4. Was receiving specific diet and exercise (if any) therapies during the observation period.

Exclusion Criteria:

1. Had taken other diabetic medications than metformin within 12 weeks before the initiation of the treatment period (Week 0).
2. With a history or symptoms of lactic acidosis.

Ages: 26 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Diabetes and Endocrine Division, Study Director — Department of Medicine, Kawasaki Medical School

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 30 investigative sites in Japan from 22 August 2008 to 28 April 2009.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with uncontrolled blood glucose despite treatment with metformin as well as diet and exercise were enrolled in one of 3, once-daily (QD), twice daily (BID) or three times daily (TID) treatment groups.
Groups:
- Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID: Alogliptin 12.5 mg, tablets, orally, once daily and metformin 250 mg, tablets, orally, twice or three times daily for up 12 weeks.
- Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID: Alogliptin 25 mg, tablets, orally, once daily and metformin 250 mg, tablets, orally, twice or three times daily for up 12 weeks.
- Metformin 500mg BID or 750mg TID: Metformin 250 mg, tablets, orally, twice or three times daily and alogliptin placebo-matching tablets, orally, once daily for up 12 weeks.
Period: Overall Study
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Started | 92 | 96 | 100
Completed | 91 | 93 | 100
Not Completed | 1 | 3 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Schedule Conflict | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID | Total
Number analyzed (Participants) | 92 | 96 | 100 | 288
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.80) | 52.3 (8.02) | 52.1 (8.05) | 52.6 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 28 | 90
  Male | 60 | 66 | 72 | 198

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Analysis based on last observation carried forward, where the last postbaseline double-blind observed value is carried forward and used for all subsequent scheduled time points where data is missing. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 92 | 96 | 100
percentage of Glycosylated Hemoglobin | -0.54 (0.562) | -0.64 (0.488) | 0.21 (0.641)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.751, 95% CI 2-sided [-0.923 to -0.579]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.858, 95% CI 2-sided [-1.019 to -0.697]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 2).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 2 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 92 | 96 | 100
percentage of Glycosylated Hemoglobin | -0.13 (0.196) | -0.13 (0.150) | 0.06 (0.197)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.191, 95% CI 2-sided [-0.247 to -0.135]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.192, 95% CI 2-sided [-0.242 to -0.143]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 92 | 96 | 100
percentage of Glycosylated Hemoglobin | -0.29 (0.279) | -0.31 (0.268) | 0.09 (0.302)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Hazard Ratio, log = -0.386, 95% CI 2-sided [-0.469 to -0.303]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.403, 95% CI 2-sided [-0.484 to -0.323]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 92 | 96 | 100
percentage of Glycosylated Hemoglobin | -0.49 (0.488) | -0.56 (0.404) | 0.13 (0.465)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.621, 95% CI 2-sided [-0.757 to -0.486]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Hazard Ratio, log = -0.692, 95% CI 2-sided [-0.814 to -0.569]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 91 | 95 | 100
mg/dL | -19.2 (21.10) | -23.2 (24.17) | 0.0 (26.37)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -19.26, 95% CI 2-sided [-26.12 to -12.40]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -23.27, 95% CI 2-sided [-30.43 to -16.12]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 91 | 96 | 100
mg/dL | -19.8 (25.28) | -23.5 (26.05) | -2.2 (23.37)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -17.60, 95% CI 2-sided [-24.54 to -10.66]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -21.35, 95% CI 2-sided [-28.32 to -14.39]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 91 | 96 | 100
mg/dL | -22.0 (23.05) | -21.3 (25.30) | -3.1 (26.23)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -18.87, 95% CI 2-sided [-25.95 to -11.79]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -18.16, 95% CI 2-sided [-25.43 to -10.90]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 or final visit and baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 91 | 96 | 100
mg/dL | -19.0 (23.23) | -23.1 (27.84) | -0.8 (32.20)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -18.24, 95% CI 2-sided [-26.32 to -10.16]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -22.38, 95% CI 2-sided [-30.87 to -13.88]

9. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 12).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 12 or final visit and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Number analyzed (Participants) | 91 | 94 | 100
mg/dL | 61.7 (43.42) | 64.2 (34.76) | 70.6 (35.31)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.89, 95% CI 2-sided [-20.14 to 2.37]
Statistical Analysis 2: Comparison: Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID vs Metformin 500mg BID or 750mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.41, 95% CI 2-sided [-16.34 to 3.52]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 30 days after receiving the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID | Metformin 500mg BID or 750mg TID
Serious Adverse Events (participants affected / at risk) | 0/92 | 2/96 | 0/100
Other Adverse Events (participants affected / at risk) | 32/92 | 37/96 | 29/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID (N=92) | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID (N=96) | Metformin 500mg BID or 750mg TID (N=100)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Metformin 500mg BID or 750mg TID (N=92) | Alogliptin 25mg QD and Metformin 500mg BID or 750mg TID (N=96) | Metformin 500mg BID or 750mg TID (N=100)
Nasopharyngitis (Infections and infestations) | 18 | 22 | 20
Headache (Nervous system disorders) | 6 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 3 | 1
Blood lactic acid increased (Investigations) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.